CLINICAL TRIAL: NCT06607211
Title: Cerebral Hypoperfusion at Transcranial Color-Coded Doppler. Effects of a Treatment Protocol in Patients With Acute Brain Injury
Brief Title: Cerebral Hypoperfusion at Transcranial Color-Coded Doppler.
Acronym: IPOPERT
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 6521
Record Dates: First submitted 2024-09-19; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Cerebral Injury
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Transcranial Color-Coded Doppler (TCCD) — As part of the clinical practice, the examination will be performed with ultrasound machines that have presets for TCCD, using a low-frequency sector probe (2-25 MHz) with a transtemporal approach to obtain a scan through the midbrain plane. Through the use of Color Doppler and Pulsed-Wave Doppler, a spectral doppler waveform of the M1 segment of the middle cerebral artery velocity is obtained bilaterally. If hypoperfusion signs are discovered, TCCD will be repeated to assess the effects of each intervention.

SUMMARY:
Background. Cerebral ischemia is a major secondary factor contributing to worsening outcomes in patients with acute brain injuries. Transcranial Color-Coded Doppler (TCCD) is a reliable method for evaluating cerebral perfusion and is recommended for use in emergency settings to reduce secondary injuries. However, there is no established treatment protocol for managing cerebral hypoperfusion as detected by TCCD.

Objective. The primary objective of this study is to assess the efficacy of individual steps in a standardized treatment protocol to normalize TCCD parameters in patients with cerebral hypoperfusion. The secondary objective is to investigate the concordance between invasive intracranial pressure (ICP) measurements and those estimated through TCCD using the Czosnyka formula.

Methods. This prospective multicenter observational study will enroll patients with acute brain injury admitted in emergency or intensive care settings. Inclusion criteria include age over 18, Glasgow Coma Scale <9, and evidence of cerebral hypoperfusion based on TCCD performed on M1 tract of at least one middle cerebral artery. The hypoperfusion is defined as the concurrent presence of at least two of the following parameters: mean velocity below 30 cm/s, diastolic velocity below 20 cm/s, pulsatility index above 1.4.

Patients will undergo a stepwise treatment approach involving normocapnia verification, autoregulation testing increasing mean arterial pressure by 10 mmHg, and hyperosmolar therapy. The effectiveness of each intervention will be assessed by TCCD readings.

Endpoints. The primary endpoint is the percentage of patients who normalize cerebral perfusion parameters at each step of the protocol. The secondary endpoint is the concordance between invasive ICP measurements and those estimated through TCCD.

Sample Size. The study aims to recruit 100 patients over 24 months. Data analysis will include descriptive statistics, with significant results considered at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Patients with intraparenchymal cerebral hemorrhage, subarachnoid hemorrhage, head trauma, or hydrocephalus
* Glasgow Coma Scale belowe 9
* Need for invasive mechanical ventilation
* Arterial catheter for invasive blood pressure monitoring and blood sampling
* Presence of Doppler parameters of cerebral hypoperfusion (concurrent presence of two or more of the following conditions: PI > 1.4, diastolic velocity < 20 cm/s, and mean velocity < 30 cm/s detected in at least one middle cerebral artery)

Exclusion Criteria:

* Absence of transtemporal windows bilaterally on TCCD
* Documented severe aortic valve insufficiency
* Heart rate less than 40 bpm
* Patients with suspected vasospasm on TCCD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients with severe acute brain injury in a coma admitted to the Emergency Department or Intensive Care Unit will be subjected to TCCD as routinely done as part of clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
TCCD normalization | 1 hour
  To assess the percentage of patients who normalize TCCD cerebral perfusion parameters at each step of the protocol

SECONDARY OUTCOMES:
ICP concordance | 1 hour
  To calculate the concordance coefficients between invasively measured ICP values and those obtained through TCCD using the Czosnyka formula

CONTACTS AND LOCATIONS:
Overall Officials: Anselmo Caricato, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, UOSD TERAPIA INTENSIVA NEUROCHIRURGICA, Rome, Lazio, Italy